CLINICAL TRIAL: NCT00004182
Title: Phase II Study for the Evaluation of CPT-11 (Irinotecan, Camptosar) in Patients With Metastatic or Recurrent Breast Cancer
Brief Title: Irinotecan in Treating Patients With Metastatic or Recurrent Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: NU 98B3; NU-98B3; P-UPJOHN-976475150; NCI-G99-1642
Record Dates: First submitted 2000-01-21; First posted 2004-08-20 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of irinotecan in treating patients who have metastatic or recurrent breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate to irinotecan in patients with metastatic breast cancer who have received prior anthracycline and taxane based chemotherapy for metastatic disease. II. Determine the toxicities of irinotecan in these patients. III. Determine survival time, duration of response, and time to treatment failure in these patients after this therapy.

OUTLINE: Patients receive irinotecan IV over 90 minutes weekly for 4 weeks. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity. Patients are followed at day 30, then every 3 months.

PROJECTED ACCRUAL: A total of 14-29 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven advanced breast cancer Must have received anthracycline and taxane based chemotherapy for metastatic disease Measurable disease No CNS metastases or carcinomatous meningitis Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Menopausal status: Not specified Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Granulocyte count greater than 1500/mm3 Hemoglobin at least 9.0 g/dL Platelet count greater than 100,000/mm3 Hepatic: Bilirubin no greater than 1.3 mg/dL SGOT no greater than 3 times upper limit of normal (no greater than 5 times ULN if liver involvement) No Gilbert's disease Renal: Creatinine no greater than 2.0 mg/dL Calcium at least 12.0 mg/dL Cardiovascular: No myocardial infarction in the past 6 months No congestive heart failure requiring therapy Other: No active or uncontrolled infection HIV negative No psychiatric disorder that would preclude study No prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix No history of seizures No uncontrolled diabetes mellitus (random blood sugar at least 200 mg) No other severe disease that would preclude study Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Greater than 4 weeks since prior chemotherapy No prior irinotecan or topotecan Endocrine therapy: Not specified Radiotherapy: Greater than 4 weeks since prior radiotherapy No radiotherapy to greater than 30% of bone marrow Surgery: Not specified Other: No concurrent phenytoin, phenobarbitol, or other antiepileptic prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10; Primary Completion 2000-04 (Actual); Study Completion 2000-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J. Gradishar, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (2):
- United States (2):
  - Stanford University Medical Center, Stanford, California
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois